CLINICAL TRIAL: NCT04827459
Title: Sleep Coach: A Mobile App to Address Insomnia Symptoms Among Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2021.004; HUM00194610 (Other: University of Michigan)
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Insomnia; Breast Cancer; Prostate Cancer; Colon Cancer
Keywords: cancer survivor
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Breast Neoplasms; Prostatic Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MI Sleep Coach Mobile Application (Experimental): The Sleep Coach app includes evidence-based CBT-I strategies, interactive activities and a computerized dialogue agent to engage users in the adoption of and adherence to CBT-I strategies.
  Interventions: Behavioral: Sleep Coach App

INTERVENTIONS:
Behavioral: Sleep Coach App — Participants will be encouraged to interact with the mobile app daily for as much time as they wish, or for as little as 5 - 10 minutes, over a 7-week period.
  Other Names: MI Sleep Coach

SUMMARY:
This clinical trial will evaluate the adherence, usefulness, satisfaction and effect size for the Sleep Coach app as an intervention for insomnia in 30 adult post-treatment cancer survivors.

DETAILED DESCRIPTION:
Difficulty sleeping, falling and/or staying asleep, is common in people after they have been diagnosed and treated for cancer. Cognitive Behavioral Therapy for Insomnia (CBT-I) is considered to be the preferred treatment but until now, there has been limited access for most people to CBT-I because it has required an in-person visit with a trained therapist. This research study is to test a mobile CBT-I app called MI Sleep Coach to deliver CBT-I. The goal of this study is to understand if people are willing to use the app, if they find it useful in helping with sleep difficulty and if they are satisfied with using it. The investigators hope to use information from this small feasibility study to study the effectiveness of the app in a larger group of cancer survivors and ultimately to help cancer survivors with sleep difficulties to sleep better.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Has completed curative-intent treatment (chemo, surgery, RT) for prostate, colon or breast cancer at least three months and not more than 5 years prior to study entry. Note: Ongoing hormonal therapy (i.e., tamoxifen, aromatase inhibitors, casodex), Herceptin and maintenance therapies are allowed.
* Ability to read and write English
* Ability to complete questionnaire(s) by themselves or with assistance.
* Reports trouble falling asleep or staying asleep on at least 3 nights per week (most weeks) for the last 3 months.
* Own an Android phone version 8 or higher (The latest version of Android is 11.0) or an iPhone running iOS 11 or higher (The latest version of iOS is 14.3.)
* Ability to provide informed written consent.

Exclusion Criteria:

* Inability to read and write English
* Diagnosis of a sleep disorder other than insomnia (e.g. sleep apnea, restless legs syndrome, narcolepsy)
* Diagnosis of Insomnia prior to cancer diagnosis
* Reports physical symptoms that interfere with sleep, such as shortness of breath, pain, hot flashes, frequent urination
* Major psychiatric or medical condition other than cancer suspected to contribute to their sleep disturbance
* Evidence of active cancer (i.e. not considered NED)
* Currently or previously received CBT-I
* Patients who are night shift workers or subject to other external restrictions on their opportunity to sleep at night.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Percentage of participants engaging with the app at least 4 days/week | 7 weeks
  Adherence will be evaluated using data gathered from the application. Participants will be asked to interact daily with the application and will be deemed adherent if they interact with the app at least 4 times per week for the duration (7 weeks) of the study. Adherence rate will be the number of participants deemed adherent / total number of participants.
Percentage of participants that find the intervention useful | 7 weeks
  Usefulness will be assessed using a survey developed by the investigators of this study called the User Experience Survey, which is based upon the Unified Theory of Acceptance and Use of Technology (UTAUT). The survey assesses perceived ease of use and usefulness of the Sleep Coach app as well as participant satisfaction with the app. To assess usefulness, participants are asked to rate the usefulness of 10 different features of the Sleep Coach app on a scale of 1 to 4, with higher scores indicating greater usefulness. Participants who rate at least one app feature 2 or greater will be considered as finding the intervention useful.
Percentage of participants satisfied with the intervention | 7 weeks
  Satisfaction will be assessed using 2 questions from the User Experience Survey: one to determine the level of overall satisfaction with the app and the other to determine the level of willingness to recommend the app to others. Satisfaction questions are rated on a scale of 1 to 5, with higher scores indicating greater agreement/satisfaction. Participants who rate both questions 4 or greater will be considered satisfied with the Sleep Coach app.

SECONDARY OUTCOMES:
Effect size of the intervention as measured by the Insomnia Severity Index (ISI). | baseline to 7 weeks
  The ISI is a 7-item questionnaire used to measure a patient's perceptions of the nature, impact and severity of insomnia. Items are scored on a scale of 0 to 4, with higher scores indicating more severe insomnia. Cohen's d or f will be calculated from baseline to week 7 to assess the effect size of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Noel Arring, DNP, PhD, RN, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arring N, Barton DL, Lafferty C, Cox B, Conroy DA, An L. Mi Sleep Coach Mobile App to Address Insomnia Symptoms Among Cancer Survivors: Single-Arm Feasibility Study. JMIR Form Res. 2024 Apr 26;8:e55402. doi: 10.2196/55402. PMID 38669678